CLINICAL TRIAL: NCT00495898
Title: A German Multicenter, Randomized, Controlled, Open-Label Study of the Cypher Sirolimus-Eluting Stent in the Treatment of Diabetic Patients With De Novo Native Coronary Artery Lesions
Brief Title: A Study of Diabetic Patients With De Novo Native Coronary Artery Lesions
Acronym: SCORPIUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRDDE-001
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CYPHER sirolimus-eluting stent
  Interventions: Device: CYPHER sirolimus-eluting stent
- 2 (Active Comparator): uncoated Bx VELOCITY balloon-expandable stent
  Interventions: Device: uncoated Bx VELOCITY balloon-expandable stent

INTERVENTIONS:
Device: CYPHER sirolimus-eluting stent — drug-eluting stent
  Arms: 1
Device: uncoated Bx VELOCITY balloon-expandable stent — bare metal stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the CYPHER sirolimus-eluting stent in maintaining minimum lumen diameter in de novo native coronary artery lesions as compared to the uncoated Bx VELOCITY balloon-expandable stent in patients with manifest diabetes mellitus. Both stents are mounted on the Raptorâ Rapid Exchange Stent Delivery System.

DETAILED DESCRIPTION:
This is a multicenter (19 sites), prospective, 2 arm randomized study designed to assess the safety and effectiveness of the CYPHER sirolimus-eluting stent as compared to the uncoated Bx VELOCITY balloon-expandable stent in patients with manifest diabetes mellitus. Patients with de novo native coronary artery lesions <= 42 mm in length and >=2.5mm and <=3.5mm in diameter (by visual estimate) will be included in the study. A total of 190 patients will be entered and randomly allocated to the CYPHERTM sirolimus-eluting stent or the uncoated Bx VELOCITY balloon-expandable stent at a 1:1 ratio. Patients will be followed for 12 months post-procedure, with all patients having a repeat angiography at 8 months (± 1 month).

It is anticipated the total duration of the study will be 18 months: 6 months to complete patient enrollment and 12 months for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B I-II) OR patients with documented silent ischemia;
* Manifest diabetes mellitus, proven by fasting glucose (12 h) > 127 mg/dl or oral glucose challenge: >= 200 mg/dl after 2 h or diabetes mellitus already treated with oral antidiabetics or insulin;
* Treatment of a de novo native coronary artery lesion in a major coronary artery in patients with single or multi-vessel disease; patients with 2- or more-vessel-disease can be enrolled if previous treatment(s) of those lesions other than the target lesion have taken place at least 3 months prior to the enrolment to this study. If more than 1 study stent is necessary to treat the lesion, overlapping is strongly recommended;
* Target vessel diameter at the lesion site is >= 2.5mm and <= 3.5mm (visual estimate); (stents will be available in 2.5 / 3.0 mm width);
* Target lesion is <= 42mm in length (visual estimate); (stents will be available in 8, 18 and 33 mm length);
* Target lesion diameter stenosis is > 50% and <100% (visual estimate);

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2002-11; Primary Completion 2005-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
angiographic in-segment late loss | 8 months post-procedure

SECONDARY OUTCOMES:
late loss | 8 months post-procedure
angiographic binary restenosis | 8 months post-procedure
target lesion revascularization (TLR) | 8 months post-procedure
target vessel revascularization (TVR) | 8 months post-procedure
target vessel failure (TVF) | 8 months post-procedure
procedure success | 8 months post-procedure
lesion success rate | 0
resource use | 1 year post-procedure
productivity loss | 1 year post-procedure
Major Adverse Cardiac Events (MACE) | 30 days, and 8 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich Baumgart, MD, PhD, Principal Investigator — Universität Duisburg-Essen
Locations (1):
- University of Essen, Essen, Germany

REFERENCES:
- [Result] Baumgart D, Klauss V, Baer F, Hartmann F, Drexler H, Motz W, Klues H, Hofmann S, Volker W, Pfannebecker T, Stoll HP, Nickenig G; SCORPIUS Study Investigators. One-year results of the SCORPIUS study: a German multicenter investigation on the effectiveness of sirolimus-eluting stents in diabetic patients. J Am Coll Cardiol. 2007 Oct 23;50(17):1627-34. doi: 10.1016/j.jacc.2007.07.035. PMID 17950142
- [Derived] Sinning JM, Baumgart D, Werner N, Klauss V, Baer FM, Hartmann F, Drexler H, Motz W, Klues H, Voelker W, Pfannebecker T, Stoll HP, Nickenig G; SCORPIUS Study. Five-year results of the Multicenter Randomized Controlled Open-Label Study of the CYPHER Sirolimus-Eluting Stent in the Treatment of Diabetic Patients with De Novo Native Coronary Artery Lesions (SCORPIUS) study: a German multicenter investigation on the effectiveness of sirolimus-eluting stents in diabetic patients. Am Heart J. 2012 Mar;163(3):446-53, 453.e1. doi: 10.1016/j.ahj.2011.12.010. PMID 22424016